CLINICAL TRIAL: NCT00307151
Title: Phase II, Parallel, Randomized, Clinical Trials Comparing the Responses to Initiation of NNRTI-Based Versus PI-Based Antiretroviral Therapy in HIV Infected Infants Who Have and Have Not Previously Received Single Dose Nevirapine for Prevention of Mother-to-Child HIV Transmission
Brief Title: Antiviral Responses to NNRTI-Based vs. PI-Based ARV Therapy in HIV Infected Infants Who Have or Have Not Received Single Dose NVP for Prevention of Mother-to-Child Transmission of HIV
Acronym: P1060
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT P1060; U01AI068632 (NIH)
Record Dates: First submitted 2006-03-24; First posted 2006-03-27 (Estimated); Results first posted 2011-08-03 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: HIV Infections
Keywords: Treatment Naive; Mother-To-Child Transmission; MTCT; Pediatrics; Viral resistance
MeSH Terms: conditions — HIV Infections | interventions — Lamivudine; Lopinavir; lopinavir-ritonavir drug combination; Nevirapine; Zidovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Coh I: NVP (Experimental): Cohort I: Previously received single dose nevirapine (SD NVP). Randomly assigned to receive an NNRTI-based regimen.
  Interventions: Drug: Lamivudine; Drug: Nevirapine; Drug: Zidovudine
- Coh I: LPV/r (Experimental): Cohort I: Previously received SD NVP. Randomly assigned to receive a PI-based regimen.
  Interventions: Drug: Lamivudine; Drug: Lopinavir/ritonavir; Drug: Zidovudine
- Coh II: NVP (Experimental): Cohort II: Did not previously receive SD NVP. Randomly assigned to receive an NNRTI-based regimen
  Interventions: Drug: Lamivudine; Drug: Nevirapine; Drug: Zidovudine
- Coh II: LPV/r (Experimental): Cohort II: Did not previously receive SD NVP. Randomly assigned to receive a PI-based regimen
  Interventions: Drug: Lamivudine; Drug: Lopinavir/ritonavir; Drug: Zidovudine

INTERVENTIONS:
Drug: Lamivudine — 4 mg/kg twice daily
  Other Names: 3TC; Epivir
Drug: Lopinavir/ritonavir — 16/4 mg/kg twice daily for participants 2 months of age to less than 6 months of age; 12/3 mg/kg twice daily for participants at least 6 months of age and weighing less than 15 kg; 10/2.5 mg/kg twice daily for participants at least 6 months of age and weighing between 15 kg and 40kg; 400/100 mg twice daily for participants weighing more than 40 kg
  Other Names: LPV/r; Kaletra; LPV/RTV
  Arms: Coh I: LPV/r; Coh II: LPV/r
Drug: Nevirapine — Initially: 4 mg/kg for 14 days, then 7 mg/kg twice daily. In protocol version 2.0, Letter of Amendment 1 (September 2007), NVP dose increased to conform with WHO guidelines to: 160 to 200 mg/m^2/dose to max 200 mg once daily for 14 days, then 160 to 200 mg/m^2/dose to max 200 mg twice daily
  Other Names: NVP; Viramune
  Arms: Coh I: NVP; Coh II: NVP
Drug: Zidovudine — 180 mg/m^2 twice daily
  Other Names: ZDV; AZT; Retrovir

SUMMARY:
A single dose of nevirapine (SD NVP) given to an HIV infected pregnant woman followed by a single dose to her infant has been shown to be an effective way of reducing the risk of mother-to-child transmission (MTCT) of HIV. The purpose of this study was to compare the effectiveness of a non-nucleoside reverse transcriptase inhibitor (NNRTI)-based antiretroviral regimen versus a protease inhibitor (PI)-based regimen in HIV infected infants who had or had not been exposed to SD NVP for prevention of MTCT.

>>

>> A five year follow up has been added to the study.

DETAILED DESCRIPTION:
Single dose nevirapine (SD NVP) has greatly reduced the rate of mother-to-child transmission (MTCT) of HIV. Non-nucleoside reverse transcriptase inhibitor (NNRTI)-based regimens are recommended for use by the World Health Organization (WHO) in resource-limited settings. However, research suggests that mothers and infants exposed to SD NVP experience higher virologic failure rates when treated with NNRTI-based regimens than their unexposed counterparts. Data show that the use of SD NVP is associated with NNRTI resistance in HIV infected women and infants. The purpose of this trial was to compare and evaluate virologic responses to an NNRTI-based regimen versus a protease-inhibitor (PI)-based regimen in HIV infected infants who had or had not been exposed to SD NVP intrapartum and after birth.

>>

>> Participants were enrolled into one of two Cohorts with proposed enrollment into each Cohort of 288 participants. Cohort I participants must have received SD NVP for prevention of MTCT. Cohort II participants and their mothers must not have previously received NVP or any other NNRTIs. Participants in both Cohorts were randomly assigned to receive either an NNRTI (Coh I:NVP and Coh II: NVP) or PI (Coh I: LPV/r and Coh II: LPV/r) -based regimen. The NNRTI-based regimen included NVP, zidovudine (ZDV) and lamivudine (3TC). The PI-based regimen included lopinavir/ritonavir (LPV/r), ZDV and 3TC. If participants experienced adverse reactions to ZDV, stavudine (d4T) could be substituted. Randomization was stratified by age (6-<12 months vs. >=12 months, with the 2-<6 month stratum added in protocol version 4.0 when the lower age limit was decreased from 6 months to 2 months).

>>

>> Study visits were scheduled at entry, weeks 2, 4, 8, 12, 16, 24 and then every 24 weeks. A physical exam, blood collection, and assessments of HIV-related symptoms occurred at all visits.

>>

>> Based on a Data Safety and Monitoring Committee (DSMB) review of study data on April 20 2009, enrollment to Cohort I was closed and interim results released. Data from this and another similar study (AIDS Clinical Trials Group (ACTG) A5208) conducted in mothers, showed that the PI-based regimen was more effective than the NNRTI-based regimen in infants who had received SD NVP for prevention of MTCT. Cohort II was allowed to remain open for enrollment and the lower age limit for enrollment reduced from 6 months to 2 months.

>>

>> In June 2010, follow-up for all subjects was extended from the original 24 weeks beyond enrollment of the last subject to 48 weeks. On October 27 2010, the DSMB conducted a final review of Cohort II data, and recommended results be unblinded and released. As found in Cohort I, the PI-based regimen was more effective than the NNRTI-based regimen in infants who had not been previously exposed to SD NVP for PMTCT. Primary and secondary outcome results for Cohort I include all follow-up until April 20, 2009 and for Cohort II, all follow-up until October 27, 2010.

>>

>> Version 5.0 of the protocol (March 21, 2011) extended follow-up on all subjects for an additional 5 years to December 2016. The purpose of the extension was to collect long term safety and virologic efficacy data in this study population and to pilot administration of a series of neuropsychological tests. During the extension, participants did not receive any medications through the study, but instead through their local clinics. Clinic visits took place every 3 months. Adverse event summaries use all follow-up in both Cohorts until December, 2016.

>>

>>

ELIGIBILITY:
Inclusion Criteria for All Participants:>>

* age >=6 months to < 36 months (decreased to 2 months in protocol version 4.0)>>
* HIV infected>>
* Viral load greater than 5,000 copies/ml within 60 days of study entry>>
* Treatment naive except for antiretrovirals (ARV) used to prevent MTCT (infant ARV use for <=1 week postpartum for prevention of MTCT allowed) >>
* Eligible for treatment according to WHO pediatric algorithm (updated in protocol version 1.0, Letter of amendment (LOA)#1) and protocol version 2.0, LOA#3). Subjects with active opportunistic infections were not eligible for study participation until they had been treated and were clinically stable >>
* Parent or legal guardian willing to provide signed informed consent>>

Inclusion Criteria for Cohort I:>>

* Documentation of maternal or infant NVP exposure or a highly reliable verbal report. (Updated in protocol version 2.0, LOA#3 to require written clinic/hospital documentation of infant exposure to SD NVP)>>
* Use of maternal ARV, including NVP, permitted during pregnancy>>
* One or more of the following: strict formula feeding, initial infant HIV diagnosis occurring while younger than 60 days of age, or an initial AIDS-defining illness diagnosis by WHO criteria while younger than 60 days of age. >>

Inclusion Criteria for Cohort II:>>

* Use of maternal ARVs, excluding NNRTIs, permitted during pregnancy>>
* Evidence of lack of prior NVP exposure (added in protocol version 2.0, LOA#3) by review of maternal and child medical records or health card (or other written documentation) for evidence of NVP exposure to mother or infant during pregnancy, labor, and delivery. If no written documentation showing lack of NVP use was shown in these records or if these records were not available for review, then a verbal report considered to be highly reliable by the study nurse was acceptable AND one or more of the following: >>

  1. Study subject born before single dose NVP was available for prevention of MTCT of HIV in the location of birth of study subject>>
  2. Study subject born before the biological mother's first positive HIV test>>
  3. Site staff had another reason to believe the subject had not been exposed to NVP >> >> Exclusion Criteria for All Participants:>>
* Grade 2 or higher aspartate aminotransferase (AST) or alanine aminotransferase (ALT) at study screening>>
* Grade 3 or higher laboratory toxicity at study screening>>
* Received ARVs for anything other than the prevention of intrapartum MTCT. Infants who received ARVs after the first week of life (e.g., for the prevention of MTCT of HIV through breastfeeding) were excluded >>
* Acute serious infections requiring active treatment. Subjects could be receiving treatment for active TB if it did not include rifamycin drugs>>
* Receiving chemotherapy for an active tumor>>
* History of a cardiac conduction abnormality and underlying structural heart disease>>
* Required certain medications>> >> Exclusion Criteria for Cohort I: >>
* History of or currently breastfeeding. Breastfed infants with a positive HIV test or who had experienced an AIDS-defining illness by WHO criteria at 60 days of age or younger were not excluded>>

Exclusion Criteria for Cohort II:>>

* Exposure to any maternal NVP or other NNRTI prior to or during the pregnancy or while breastfeeding>>
* Exposure of infant to NVP at any time including during the first week of life

Ages: 2 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 452 (Actual)
Dates: Start 2005-12; Primary Completion 2010-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Palumbo, MD, Study Chair — Division of Infectious Diseases and International Health, Dartmouth-Hitchcock Medical Center; Avy Violari, MD, Study Chair — Perinatal HIV Research Unit, University of Witwatersrand
Locations (10):
- BJ Medical College CRS, Pune, Maharashtra, India
- University of North Carolina Lilongwe CRS, Mzimba Road, Lilongwe, Malawi
- South Africa (4):
  - Nelson R. Mandela School of Medicine, University of Kwazulu, Natal, Durban
  - University of Stellenbosch-Tygerberg Hospital, South Africa, Cape Town
  - Harriet Shezi Clinic at Chris Hani Baragwanath Hospital, Johannesburg
  - Perinatal HIV Research Unit, Chris Hani Baragwanath Hospital, Johannesburg
- Kilimanjaro Christian Medical CRS, IDC Research Offices, Moshi, Tanzania
- Makerere University, Kampala, Uganda
- George Clinic CRS, Lusaka, Zambia
- UZ-College of Health Sciences, Harare, Zimbabwe

REFERENCES:
- [Background] Arrive E, Newell ML, Ekouevi DK, Chaix ML, Thiebaut R, Masquelier B, Leroy V, Perre PV, Rouzioux C, Dabis F; Ghent Group on HIV in Women and Children. Prevalence of resistance to nevirapine in mothers and children after single-dose exposure to prevent vertical transmission of HIV-1: a meta-analysis. Int J Epidemiol. 2007 Oct;36(5):1009-21. doi: 10.1093/ije/dym104. Epub 2007 May 28. PMID 17533166
- [Background] Chi BH, Sinkala M, Stringer EM, Cantrell RA, Mtonga V, Bulterys M, Zulu I, Kankasa C, Wilfert C, Weidle PJ, Vermund SH, Stringer JS. Early clinical and immune response to NNRTI-based antiretroviral therapy among women with prior exposure to single-dose nevirapine. AIDS. 2007 May 11;21(8):957-64. doi: 10.1097/QAD.0b013e32810996b2. PMID 17457089
- [Background] Eshleman SH, Hoover DR, Hudelson SE, Chen S, Fiscus SA, Piwowar-Manning E, Jackson JB, Kumwenda NI, Taha TE. Development of nevirapine resistance in infants is reduced by use of infant-only single-dose nevirapine plus zidovudine postexposure prophylaxis for the prevention of mother-to-child transmission of HIV-1. J Infect Dis. 2006 Feb 15;193(4):479-81. doi: 10.1086/499967. Epub 2006 Jan 11. PMID 16425125
- [Background] White PD. What causes prolonged fatigue after infectious mononucleosis: and does it tell us anything about chronic fatigue syndrome? J Infect Dis. 2007 Jul 1;196(1):4-5. doi: 10.1086/518615. Epub 2007 May 24. No abstract available. PMID 17538875
- [Background] Sankatsing RR, Wit FW, Pakker N, Vyankandondera J, Mmiro F, Okong P, Kastelein JJ, Lange JM, Stroes ES, Reiss P. Effects of nevirapine, compared with lamivudine, on lipids and lipoproteins in HIV-1-uninfected newborns: the stopping infection from mother-to-child via breast-feeding in Africa lipid substudy. J Infect Dis. 2007 Jul 1;196(1):15-22. doi: 10.1086/518248. Epub 2007 May 16. PMID 17538878
- [Result] Palumbo P, Lindsey JC, Hughes MD, Cotton MF, Bobat R, Meyers T, Bwakura-Dangarembizi M, Chi BH, Musoke P, Kamthunzi P, Schimana W, Purdue L, Eshleman SH, Abrams EJ, Millar L, Petzold E, Mofenson LM, Jean-Philippe P, Violari A. Antiretroviral treatment for children with peripartum nevirapine exposure. N Engl J Med. 2010 Oct 14;363(16):1510-20. doi: 10.1056/NEJMoa1000931. PMID 20942667
- [Result] Palumbo P, Violari A, Lindsey J, Hughes M, Jean-Philippe P, Mofenson L, Purdue L, Eshleman S for the IMPAACT P1060 Study Team. Nevirapine vs Lopinavir-ritonavir-based antiretroviral therapy in single dose Nevirapine-exposed HIV-infected infants: preliminary results from the IMPAACT P1060 Trial. 5th IAS Conference on HIV Pathogenesis, Treatment and Prevention, Capetown, July, 2009.
- [Result] Palumbo P, Violari A, Lindsey J, Hughes M, Jean-Philippe P, Mofenson L, Bwakura-Dangarembizi M, Kamthunzi P, Eshleman S and Prudue L for the IMPAACT P1060 Team. Nevirapine (NVP)-vs. Lopinavir-Ritonavir (LPV/r)-based antiretroviral therapy (ART) among HIV-infected infants in resource-limited settings: The IMPAACT P1060 Trial. 18th Conference on Retroviruses and Opportunistic Infections, Boston, February, 2011.
- [Derived] Patel K, Lindsey J, Angelidou K, Aldrovandi G, Palumbo P; IMPAACT P1060 Study Team. Metabolic effects of initiating lopinavir/ritonavir-based regimens among young children. AIDS. 2018 Oct 23;32(16):2327-2336. doi: 10.1097/QAD.0000000000001980. PMID 30102656
- [Derived] Angelidou K, Palumbo P, Lindsey J, Violary A, Archary M, Barlow L, Claggett B, Hughes M, Wei LJ; International Maternal Pediatric Adolescent AIDS Clinical Trials Group (IMPAACT) P1060 Study Team. Defining Study Outcomes That Better Reflect Individual Response to Treatment. Pediatr Infect Dis J. 2018 Mar;37(3):258-262. doi: 10.1097/INF.0000000000001766. PMID 29189677
- [Derived] Barlow-Mosha L, Angelidou K, Lindsey J, Archary M, Cotton M, Dittmer S, Fairlie L, Kabugho E, Kamthunzi P, Kinikar A, Mbengeranwa T, Msuya L, Sambo P, Patel K, Barr E, Jean-Phillipe P, Violari A, Mofenson L, Palumbo P, Chi BH. Nevirapine- Versus Lopinavir/Ritonavir-Based Antiretroviral Therapy in HIV-Infected Infants and Young Children: Long-term Follow-up of the IMPAACT P1060 Randomized Trial. Clin Infect Dis. 2016 Oct 15;63(8):1113-1121. doi: 10.1093/cid/ciw488. Epub 2016 Jul 20. PMID 27439527
- [Derived] Lindsey JC, Hughes MD, Violari A, Eshleman SH, Abrams EJ, Bwakura-Dangarembizi M, Barlow-Mosha L, Kamthunzi P, Sambo PM, Cotton MF, Moultrie H, Khadse S, Schimana W, Bobat R, Zimmer B, Petzold E, Mofenson LM, Jean-Philippe P, Palumbo P; P1060 Study Team. Predictors of virologic and clinical response to nevirapine versus lopinavir/ritonavir-based antiretroviral therapy in young children with and without prior nevirapine exposure for the prevention of mother-to-child HIV transmission. Pediatr Infect Dis J. 2014 Aug;33(8):846-54. doi: 10.1097/INF.0000000000000337. PMID 25222305
- [Derived] Violari A, Lindsey JC, Hughes MD, Mujuru HA, Barlow-Mosha L, Kamthunzi P, Chi BH, Cotton MF, Moultrie H, Khadse S, Schimana W, Bobat R, Purdue L, Eshleman SH, Abrams EJ, Millar L, Petzold E, Mofenson LM, Jean-Philippe P, Palumbo P. Nevirapine versus ritonavir-boosted lopinavir for HIV-infected children. N Engl J Med. 2012 Jun 21;366(25):2380-9. doi: 10.1056/NEJMoa1113249. PMID 22716976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited at 10 study sites, 4 in South Africa and 1 each in Uganda, Zimbabwe, Zambia, Malawi, Tanzania and India between November 9, 2006 and March 19, 2010.
Pre-assignment Details: Infants and children 6 - 36 months of age (lower age limit changed to 2 months in Protocol Version 4.0) were stratified by age (2-<6 months, 6-<12 months and >=12 months) and randomly assigned to receive either AZT/3TC/NVP or AZT/3TC/LPV/r. One subject was randomized but never started study treatment.
Period: Overall Study
Arm/Group | Coh I: NVP | Coh I: LPV/r | Coh II: NVP | Coh II: LPV/r
Started | 82 | 82 | 147 | 140 (One participant never started treatment, were not followed and not included in analysis.)
Completed | 71 (Results are through date DSMB closed Cohort I to accrual (April 20, 2009)) | 75 (Results are through date DSMB closed Cohort I to accrual (April 20, 2009)) | 127 (Results are through date DSMB recommended Cohort II results be unblinded (October 27, 2010)) | 129 (Results are through date DSMB recommended Cohort II results be unblinded (October 27, 2010))
Not Completed | 11 | 7 | 20 | 11
Not completed — Death | 4 | 3 | 10 | 3
Not completed — Severe debilitation, unable to continue | 1 | 0 | 0 | 0
Not completed — Subject unable to get to clinic | 1 | 0 | 6 | 2
Not completed — Withdrew consent | 0 | 1 | 1 | 3
Not completed — Not willing to adhere to study reqs | 2 | 0 | 2 | 2
Not completed — Clinic unable to contact subject | 3 | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coh I: NVP | Coh I: LPV/r | Coh II: NVP | Coh II: LPV/r | Total
Number analyzed (Participants) | 82 | 82 | 147 | 140 | 451
Age, Customized [Number; unit: participants]
  <12 months | 60 | 63 | 41 | 36 | 200
  >=12 months | 22 | 19 | 106 | 104 | 251
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 41 | 78 | 72 | 237
  Male | 36 | 41 | 69 | 68 | 214
Race/Ethnicity, Customized [Number; unit: participants]
  Black African | 81 | 81 | 132 | 134 | 428
  Coloured | 1 | 1 | 1 | 2 | 5
  Native of India | 0 | 0 | 12 | 4 | 16
  Not available | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Tanzania | 2 | 0 | 8 | 7 | 17
  Zambia | 2 | 4 | 14 | 18 | 38
  Uganda | 1 | 4 | 20 | 20 | 45
  Malawi | 2 | 0 | 16 | 20 | 38
  South Africa | 71 | 65 | 41 | 36 | 213
  Zimbabwe | 4 | 9 | 36 | 35 | 84
  India | 0 | 0 | 12 | 4 | 16
Ever breastfed [Number; unit: participants]
  Yes | 15 | 19 | 118 | 115 | 267
  No | 67 | 63 | 29 | 25 | 184
Documentation of SD NVP use at birth [Number; unit: participants]
  Born before NVP available/mother known to have HIV | 0 | 0 | 116 | 104 | 220
  Medical record review | 62 | 63 | 10 | 12 | 147
  Verbal evidence only | 20 | 19 | 19 | 22 | 80
  Found to have received SD NVP | 0 | 0 | 2 | 2 | 4
WHO Stage [Number; unit: participants] — World Health Organization (WHO) staging system for HIV infection and disease.
  participants
    I | 7 | 18 | 29 | 25 | 79
    II | 23 | 22 | 26 | 27 | 98
    III | 39 | 38 | 80 | 77 | 234
    IV | 13 | 4 | 12 | 11 | 40
HIV-1 RNA [Number; unit: participants]
  <100,000 copies/ml | 6 | 5 | 20 | 27 | 58
  100,000 - < 750,000 copies/ml | 27 | 34 | 70 | 53 | 184
  >=750,000 copies/ml | 49 | 43 | 57 | 60 | 209
CD4 Percent [Number; unit: participants]
  <15 Percent | 24 | 21 | 73 | 69 | 187
  15 Percent - < 25 Percent | 37 | 37 | 60 | 54 | 188
  >= 25 Percent | 21 | 24 | 13 | 17 | 75
  Missing | 0 | 0 | 1 | 0 | 1
NVP resistance [Number; unit: participants]
  Yes | 7 | 11 | 1 | 4 | 23
  No | 68 | 62 | 110 | 91 | 331
  Not available | 7 | 9 | 36 | 45 | 97

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Treatment Failure, Defined as a Confirmed Virologic Failure or Permanent Discontinuation of the Randomized NNRTI or PI Component of Study Treatment
Description: Treatment failure is defined as a confirmed plasma HIV-1 RNA level that is <1 log10 copies/mL below the study entry value at 12 to 24 weeks after treatment is initiated OR a confirmed plasma HIV-1 RNA level >400 copies/mL at 24 weeks OR permanent discontinuation of the randomized NNRTI or PI component of study treatment at or prior to 24 weeks of treatment for any reason including death. Results report percent of participants reaching a treatment failure endpoint by week 24 calculated using the Kaplan-Meier method.
Time Frame: Earlier of 24 weeks or date of DSMB decision to unblind Cohort results (Coh I: April 20, 2009; Coh II: October 27, 2010)
Population: Analysis uses intent to treat population
Measure: Number; unit: Percent of participants
Arm/Group | Coh I: NVP | Coh I: LPV/r | Coh II: NVP | Coh II: LPV/r
Number analyzed (Participants) | 82 | 82 | 147 | 140
Percent of participants | 39.6 | 21.7 | 40.8 | 19.3
Statistical Analysis 1: Comparison: Coh I: NVP vs Coh I: LPV/r; Test type: Superiority or Other; p = 0.015, t-test, 2 sided — P-value not adjusted for multiple interim analyses, but adjustment would be negligible because Peto-Haybittle spending function used as basis for calculating repeated confidence intervals used in interim monitoring; Risk difference estimate stratified by age (<12 months vs. >=12 months)and reports rate on NVP arm minus rate on LPV/r arm; Risk Difference (RD) = 18.6, 95% CI 2-sided [3.7 to 33.6] — Endpoint rates with standard errors calculated from Kaplan-Meier curves for each treatment group and age stratum. Differences in week 24 failure proportions by treatment calculated weighted by the inverse of the variance in each age stratum
Statistical Analysis 2: Comparison: Coh II: NVP vs Coh II: LPV/r; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Risk difference estimate stratified by age (<12 months vs. >=12 months) and reports rate on NVP arm minus rate on LPV/r arm; Risk Difference (RD) = 21.5, 95% CI 2-sided [11.2 to 31.8] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Time From Randomization to Treatment Failure, Defined as Virologic Failure or Permanent Discontinuation of the Randomized NNRTI or PI Component of Study Treatment
Description: Treatment failure is defined as a confirmed plasma HIV-1 RNA level that is <1 log10 copies/mL below the study entry value at 12 to 24 weeks after treatment is initiated OR a confirmed plasma HIV-1 RNA level >400 copies/mL at 24 weeks OR a confirmed viral rebound >4000 copies/mL after week 24 OR permanent discontinuation of the randomized NNRTI or PI component of study treatment for any reason including death.
Time Frame: Until date of DSMB decision to unblind Cohort results (Coh I: April 20, 2009 - median follow-up 48 weeks and range 0 - 125 weeks; Coh II: October 27, 2010 - median follow-up 72 weeks and range from 0 to 204 weeks)
Population: Analysis uses intent to treat population
Measure: Number (95% Confidence Interval); unit: Weeks
Arm/Group | Coh I: NVP | Coh I: LPV/r | Coh II: NVP | Coh II: LPV/r
Number analyzed (Participants) | 82 | 82 | 147 | 140
Weeks
  10th percentile | 12 [4 to 12] | 4 [4 to 16] | 4 [2 to 8] | 14 [8 to 24]
  25th percentile | 16 [12 to 24] | 36 [16 to NA] — Not estimable as upper limit for survival function at all weeks is above 75% | 16 [12 to 24] | 36 [24 to 108]

3. Secondary Outcome: Percent of Participants Experiencing Virologic Failure
Description: Virologic failure is defined as a confirmed plasma HIV-1 RNA level that is <1 log10 copies/mL below the study entry value at 12 to 24 weeks after treatment is initiated OR a confirmed plasma HIV-1 RNA level >400 copies/mL at 24 weeks OR death on or before 24 weeks. Results report percent of participants reaching a virologic failure endpoint by week 24 calculated using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: Analysis uses intent to treat population.
Measure: Number; unit: Percent of participants
Arm/Group | Coh I: NVP | Coh I: LPV/r | Coh II: NVP | Coh II: LPV/r
Number analyzed (Participants) | 82 | 82 | 147 | 140
Percent of participants | 27.4 | 10.4 | 28.6 | 12.9

4. Secondary Outcome: Time From Randomization to Virologic Failure
Description: Virologic failure is defined as the earlier of a confirmed plasma HIV-1 RNA level that is <1 log10 copies/mL below the study entry value at 12 to 24 weeks after treatment is initiated OR a confirmed plasma HIV-1 RNA level >400 copies/mL at 24 weeks OR a confirmed viral rebound >4000 copies/mL after week 24 OR death.
Time Frame: as for outcome 2
Population: Analysis uses intent to treat population
Measure: Number (95% Confidence Interval); unit: Weeks
Arm/Group | Coh I: NVP | Coh I: LPV/r | Coh II: NVP | Coh II: LPV/r
Number analyzed (Participants) | 82 | 82 | 147 | 140
Weeks
  5th percentile | 12 [4 to 12] | 16 [2 to 24] | 12 [2 to 16] | 16 [12 to 24]
  10th percentile | 12 [12 to 24] | 24 [12 to NA] — Not estimable as upper limit for survival function at all weeks above 90% | 16 [12 to 24] | 24 [16 to 36]

5. Secondary Outcome: Time From Start of Study Treatment to First New Grade >=3 Lab Abnormality, Sign or Symptom Occurring on Study Treatment
Description: Safety events include lab abnormalities, signs or symptoms of grade 3 or higher. Events were graded according to the Division of AIDS Table for Grading Severity of Adult and Pediatric Adverse Events, Version 1.0. Events defined as new if first occurrence was after initiation of study treatment or if severity increased from entry and while on the NNRTI or PI component of study treatment.
Time Frame: On randomized NNRTI or PI component of study treatment and until date of DSMB decision to unblind Cohort results (Coh I: April 20, 2009; Coh II: October 27, 2010)
Population: Uses follow-up from start of NVP or LPV/r component of study treatment until component switched or date of DSMB decision to unblind results, whichever occurred first
Measure: Number (95% Confidence Interval); unit: Weeks
Arm/Group | Coh I: NVP | Coh I: LPV/r | Coh II: NVP | Coh II: LPV/r
Number analyzed (Participants) | 82 | 82 | 147 | 140
Weeks
  10th percentile | 4 [2 to 12] | 8 [2 to 25] | 3 [1 to 4] | 4 [2 to 5]
  25th percentile | 24 [12 to NA] — Not estimable as upper limit for survival function at all weeks above 75% | 36 [14 to 86] | 4 [4 to 6] | 12 [7 to 24]

6. Secondary Outcome: Number of Participants Developing New NRTI, NNRTI or PI-resistant Virus
Description: Numbers of participants developing new NRTI, NNRTI or PI-resistant virus after reaching a virologic failure endpoint
Time Frame: as for outcome 2
Population: Results included for any participant who was a virologic failure as defined in secondary outcome 4 and who had results available at study entry and virologic failure.
Measure: Number; unit: participants
Arm/Group | Coh I: NVP | Coh I: LPV/r | Coh II: NVP | Coh II: LPV/r
Number analyzed (Participants) | 19 | 5 | 18 | 7
participants | 16 | 1 | 10 | 4

7. Secondary Outcome: Change in CD4 Percent From Entry to Week 48
Description: Change was calculated as CD4 percent at week 48 minus entry CD4 percent (last CD4 percent before randomization date). Only subjects who reached 48 weeks of follow-up before DSMB decisions to unblind each Cohort were included in summary.
Time Frame: 48 weeks if before date of DSMB decision to unblind Cohort results (Coh I: April 20, 2009; Coh II: October 27, 2010)
Population: Analysis uses intent to treat population. Change reported if subject followed at least 48 weeks before DSMB unblinding of results for each Cohort
Measure: Mean (95% Confidence Interval); unit: Percent of CD4
Arm/Group | Coh I: NVP | Coh I: LPV/r | Coh II: NVP | Coh II: LPV/r
Number analyzed (Participants) | 63 | 70 | 109 | 119
Percent of CD4 | 13.9 [11.6 to 16.2] | 12.0 [10.3 to 13.7] | 15.2 [13.6 to 16.9] | 14.3 [13.0 to 15.7]

8. Secondary Outcome: Time From Randomization to HIV-related Disease Progression or Death
Description: HIV-related disease progression was defined as progression in WHO clinical stage from stage at entry or death. For subjects in WHO Stage IV at entry, disease progression was defined as death.
Time Frame: as for outcome 2
Population: Analysis uses intent to treat population
Measure: Number (95% Confidence Interval); unit: Weeks
Arm/Group | Coh I: NVP | Coh I: LPV/r | Coh II: NVP | Coh II: LPV/r
Number analyzed (Participants) | 82 | 82 | 147 | 140
Weeks
  5th percentile | 11 [2 to 24] | 2 [2 to 4] | 8 [2 to 24] | 35 [2 to 132]
  10th percentile | 17 [5 to NA] — Not estimable as upper limit of survival function at all weeks above 90% | 4 [2 to 24] | 35 [8 to NA] — Not estimable as upper limit of survival function at all weeks above 98% | 132 [35 to NA] — Not estimable as upper limit of survival function at all weeks above 98%

9. Secondary Outcome: Time From Randomization to Death
Description: Results report 2nd percentile of time from randomization to death
Time Frame: as for outcome 2
Population: Analysis uses intent to treat population
Measure: Number (95% Confidence Interval); unit: Weeks
Arm/Group | Coh I: NVP | Coh I: LPV/r | Coh II: NVP | Coh II: LPV/r
Number analyzed (Participants) | 82 | 82 | 147 | 140
Weeks | 11 [3 to 68] | 3 [2 to NA] — Not estimable as upper limit for survival function at all weeks above 98% | 2 [2 to 12] | 83 [3 to NA] — Not estimable as upper limit for survival function at all weeks above 98%

ADVERSE EVENTS:
Time Frame: From study enrollment until study completion
Description: Expedited adverse event (AE) reporting followed Intensive Division of AIDS (DAIDS) Reporting Level, which included AEs resulting in death, congenital anomalies, fetal losses, significant disabilities requiring hospitalization and >=grade 3 AEs defined by the "DAIDS Table for Grading the Severity of Adult and Pediatric AEs", V1.0, 12/2004.
Groups:
- Coh I: NVP: Cohort II: Previously received single dose nevirapine (SD NVP). Randomly assigned to receive an NNRTI-based regimen.
- Coh I: LPV/r: Cohort II: Previously received SD NVP. Randomly assigned to receive a PI-based regimen.
Arm/Group | Coh I: NVP | Coh I: LPV/r | Coh II: NVP | Coh II: LPV/r
All-Cause Mortality (participants affected / at risk) | 6/82 | 3/82 | 10/147 | 6/140
Serious Adverse Events (participants affected / at risk) | 23/82 | 19/82 | 65/147 | 47/140
Other Adverse Events (participants affected / at risk) | 81/82 | 82/82 | 146/147 | 140/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Coh I: NVP (N=82) | Coh I: LPV/r (N=82) | Coh II: NVP (N=147) | Coh II: LPV/r (N=140)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 5
Neutropenia (Blood and lymphatic system disorders) | 12 | 11 | 24 | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 2 | 2 | 2 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Immunosuppression (Immune system disorders) | 0 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 2 | 3
Hepatitis A (Infections and infestations) | 0 | 0 | 1 | 0
Malaria (Infections and infestations) | 0 | 0 | 6 | 6
Measles (Infections and infestations) | 0 | 0 | 1 | 1
Meningitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 10 | 6
Sepsis (Infections and infestations) | 2 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase abnormal (Investigations) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 4 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 1 | 2
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 1
Neutrophil count (Investigations) | 1 | 1 | 2 | 1
Neutrophil count decreased (Investigations) | 1 | 1 | 9 | 3
Transaminases increased (Investigations) | 1 | 0 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Hypocalcaemic seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Breath holding (Psychiatric disorders) | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Coh I: NVP (N=82) | Coh I: LPV/r (N=82) | Coh II: NVP (N=147) | Coh II: LPV/r (N=140)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 9 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 3 | 17 | 13
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 2 | 19 | 16
Neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 18 | 16
Otorrhoea (Ear and labyrinth disorders) | 3 | 0 | 12 | 4
Eye discharge (Eye disorders) | 2 | 3 | 19 | 13
Eye pruritus (Eye disorders) | 0 | 0 | 8 | 3
Ocular hyperaemia (Eye disorders) | 1 | 3 | 19 | 20
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 16 | 13
Aphthous ulcer (Gastrointestinal disorders) | 1 | 4 | 7 | 12
Diarrhoea (Gastrointestinal disorders) | 13 | 16 | 50 | 47
Stomatitis (Gastrointestinal disorders) | 1 | 3 | 8 | 12
Vomiting (Gastrointestinal disorders) | 7 | 6 | 46 | 33
Peripheral swelling (General disorders) | 2 | 1 | 5 | 8
Pyrexia (General disorders) | 13 | 17 | 68 | 68
Acarodermatitis (Infections and infestations) | 16 | 16 | 14 | 13
Body tinea (Infections and infestations) | 12 | 10 | 33 | 31
Bronchiolitis (Infections and infestations) | 4 | 5 | 12 | 8
Bronchitis (Infections and infestations) | 9 | 11 | 11 | 10
Cellulitis (Infections and infestations) | 5 | 3 | 6 | 6
Conjunctivitis (Infections and infestations) | 7 | 13 | 50 | 42
Gastroenteritis (Infections and infestations) | 20 | 23 | 31 | 24
Impetigo (Infections and infestations) | 17 | 21 | 26 | 20
Malaria (Infections and infestations) | 5 | 5 | 33 | 45
Measles (Infections and infestations) | 0 | 4 | 11 | 2
Molluscum contagiosum (Infections and infestations) | 4 | 5 | 4 | 5
Oral candidiasis (Infections and infestations) | 21 | 20 | 32 | 22
Oral herpes (Infections and infestations) | 7 | 2 | 18 | 11
Otitis externa (Infections and infestations) | 5 | 0 | 12 | 11
Otitis media (Infections and infestations) | 15 | 17 | 38 | 27
Otitis media acute (Infections and infestations) | 14 | 9 | 25 | 10
Parotitis (Infections and infestations) | 2 | 0 | 5 | 8
Persistent generalised lymphadenopathy (Infections and infestations) | 1 | 3 | 15 | 16
Pharyngitis (Infections and infestations) | 17 | 14 | 32 | 25
Plasmodium falciparum infection (Infections and infestations) | 3 | 3 | 34 | 39
Pneumonia (Infections and infestations) | 18 | 19 | 42 | 34
Pneumonia bacterial (Infections and infestations) | 2 | 11 | 27 | 22
Pulmonary tuberculosis (Infections and infestations) | 12 | 15 | 15 | 5
Purulent discharge (Infections and infestations) | 1 | 1 | 7 | 8
Subcutaneous abscess (Infections and infestations) | 2 | 5 | 3 | 6
Tinea capitis (Infections and infestations) | 19 | 33 | 55 | 54
Tinea faciei (Infections and infestations) | 8 | 1 | 8 | 6
Tinea infection (Infections and infestations) | 12 | 11 | 29 | 20
Tonsillitis (Infections and infestations) | 19 | 19 | 27 | 27
Varicella (Infections and infestations) | 7 | 9 | 13 | 9
Alanine aminotransferase (Investigations) | 9 | 4 | 21 | 8
Alanine aminotransferase increased (Investigations) | 44 | 34 | 62 | 43
Aspartate aminotransferase (Investigations) | 7 | 5 | 13 | 6
Aspartate aminotransferase increased (Investigations) | 51 | 39 | 58 | 54
Blood cholesterol increased (Investigations) | 3 | 11 | 11 | 14
Blood triglycerides increased (Investigations) | 1 | 6 | 8 | 4
Haemoglobin decreased (Investigations) | 57 | 60 | 126 | 113
Neutrophil count decreased (Investigations) | 54 | 54 | 105 | 113
Platelet count decreased (Investigations) | 3 | 8 | 19 | 23
Weight decreased (Investigations) | 2 | 5 | 18 | 21
Decreased appetite (Metabolism and nutrition disorders) | 2 | 9 | 32 | 36
Failure to thrive (Metabolism and nutrition disorders) | 7 | 11 | 13 | 8
Kwashiorkor (Metabolism and nutrition disorders) | 5 | 0 | 5 | 4
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 8 | 6
Headache (Nervous system disorders) | 2 | 0 | 10 | 10
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 8 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 14 | 61 | 60
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 13 | 7
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 9 | 7
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 22 | 20
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 9 | 52 | 48
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 10 | 9
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 6 | 10
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 | 2 | 17 | 6
Eczema (Skin and subcutaneous tissue disorders) | 10 | 10 | 20 | 15
Papule (Skin and subcutaneous tissue disorders) | 1 | 4 | 17 | 32
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 13 | 15
Rash (Skin and subcutaneous tissue disorders) | 24 | 31 | 86 | 72
Rash generalised (Skin and subcutaneous tissue disorders) | 11 | 6 | 28 | 13
Rash papular (Skin and subcutaneous tissue disorders) | 8 | 8 | 29 | 42
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 11 | 14 | 7 | 8
Skin lesion (Skin and subcutaneous tissue disorders) | 5 | 6 | 18 | 20
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 8
Skin reaction (Skin and subcutaneous tissue disorders) | 4 | 0 | 8 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 5 | 16 | 19
Swelling face (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 7
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 8 | 1
Pallor (Vascular disorders) | 1 | 0 | 8 | 1

LIMITATIONS AND CAVEATS:
Accrual to Cohort I was terminated early by the Data Safety Monitoring Committee after enrollment of 164 of the planned 288 subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trial Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscript and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.